CLINICAL TRIAL: NCT03489161
Title: The Utilization of Buprenorphine in the Emergency Room to Treat Clinical Opioid Withdrawal
Brief Title: Feasibility of the Utilization of Buprenorphine in the Emergency Room to Treat Clinical Opioid Withdrawal
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20012543
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Drug Overdose; Opioid Withdrawal; Opioid-use Disorder
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Buprenorphine (Experimental): Buprenorphine administered in the emergency room after patients presenting to the emergency department (ED) due to opioid OD who have been treated with opioid antagonist (naloxone) and are stable and alert.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — buprenorphine/naloxone 4mg/1 mg for Clinical Opioid Withdrawal Scale (COWS) scores between 8 and 12, or 8mg/2mg S/L ≥ 12 by the sublingual route

SUMMARY:
The investigators are trying to determine whether they can effectively treat patients suffering from acute opioid withdrawal in the Emergency Department at Virginia Commonwealth University Health System (VCUHS) and subsequently transfer them to an outpatient addiction clinic within the existing infrastructure. This will be a descriptive investigation of the process to reveal areas of success and opportunities for improvement in order to determine feasibility of the study procedures in preparation for a larger clinical investigation.

DETAILED DESCRIPTION:
Currently, patients in the Emergency Department at VCUHS experiencing opioid withdrawal, after reversal of opioid intoxication by naloxone, do not receive any direct treatment to stop the symptoms. They do receive indirect treatment aimed at each specific symptom, such as an anti-emetic to stop vomiting. The investigators propose directly treating all of the symptoms with the medication Suboxone, (buprenorphine/naloxone). Buprenorphine is a partial agonist on the Mu-receptor, which means it will provide less opioid effect than morphine, but should provide enough to make opioid withdrawal more tolerable. This is very important because stopping the withdrawal symptoms early will prevent the patient from quickly leaving and using opioids again, continuing their addiction cycle. The naloxone is included with buprenorphine as a deterrent to prevent intravenous injection of the drug for abuse. The investigators believe that if the patient is treated with Suboxone for withdrawal in the emergency department, and transported to the outpatient addiction treatment center at VCU, called the MOTIVATE clinic, the investigators can potentially break that cycle and help the patient work toward recovering. If successful, the investigators hope to improve the quality of life, prevent further overdose and death in those suffering from this deadly addiction.

Buprenorphine effectively treats the opioid withdrawal state. This has been demonstrated in many studies during the initial induction period with buprenorphine. Many of these patients are experiencing opioid withdrawal during this time. The sublingual dose can effectively be increased to resolve symptoms. According to many protocols and guidelines, acute opioid withdrawal is the preferred state of the patient when buprenorphine should be started.

ELIGIBILITY:
Inclusion Criteria:

* Opioid overdose only, of any formulation or route, with complete reversal of toxicity after naloxone by any route.
* RR ≥ 12
* Pulse oximetry > 95%
* GCS 15
* Clinical Opioid Withdrawal Scale (COWS) score ≥ 8

Exclusion Criteria:

* Pregnancy
* Prisoner
* Incomplete reversal of toxicity related to metrics above
* Police custody
* Known allergy to buprenorphine
* Emergent psychiatric condition including active suicidality that requires admission
* Emergent medical condition that requires admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Baseline
  Percentage of eligible potential participants who enroll in study
Acceptability of transferral to outpatient clinic (MOTIVATE) | 48 hours
  Percentage of eligible participants who complete additional screenings at MOTIVATE

SECONDARY OUTCOMES:
Feasibility of 5-Trial Delay Discounting | Prior to drug administration (within 2 hours after participant is stabilized and consented)
  Percentage of consented participants who complete this task, a brief (less than 1 minute) computer based task used to measure an individual's discounting rate when they are presented with the possibility of receiving a real reward

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States